CLINICAL TRIAL: NCT05487521
Title: Evaluation of Sleep EEG Changes in Paediatric Patients With Language Dysfunction: A Follow up Study. Evaluation of Sleep EEG Changes in Paediatric Patients With Language Dysfunction: A Follow up Study. Evaluation of Sleep EEG Changes in Pediatric Patients With Language Dysfunction : A Follow up Study
Brief Title: EEG Changes in Pediatrics With Language Dysfunction Evaluation of Sleep EEG Changes in Paediatric Patients With Language Dysfunction: A Follow up Study. EEG Changes in Pediatrics With Language Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omnia Alaa Mahsoub Abdelsalam, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: M.D4312020
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Language Disorders in Children
MeSH Terms: interventions — Methylprednisolone; Prednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patients without EEG changes or clinical seizures (No Intervention)
- Patients with EEG changes or clinical seizures (Experimental)
  Interventions: Drug: Methylprednisolone and or prednisolone

INTERVENTIONS:
Drug: Methylprednisolone and or prednisolone — we gave methylprednisolone and or prednisolone to patients with EEG activity and follow up the effect of the drug on language
  Arms: Patients with EEG changes or clinical seizures

SUMMARY:
In general, the severity of the patients' language disorders fluctuated with the degree of EEG epileptiform activity . Since then, a spectrum of disorders, often referred to collectively as the epilepsy-aphasia spectrum, have been described that share features of sleep potentiated EEG abnormalities, cognitive problems, and rare or even absent clinical seizures .

In our study , Investigators evaluated the sleep EEG changes in pediatrics with languague dysfunction then in patients with EEG changes , investigators gave treatment according to type of EEG changes and investigators did a follow up assessment of language , EEG changes and frequency of clinical seizures if present at first .

DETAILED DESCRIPTION:
Language dysfunction is one of the most common problems in paediatrics. There is increased interest in association of epilepsy and epileptiform EEG abnormalities to language dysfunction.

Electrographic status epilepticus in sleep or continuous spike - wave in slow wave during sleep, is a typical feature of acquired epileptic aphasia feature in sleep, or continuous spike-wave in slow-wave sleep, is a typical.

Our study screened for sleep potentiated epileptiform discharges in children with language dysfunction and effect of treatment of these epileptiform discharges on language dysfunction improvement.

The aim of our work :

* The primary aim of this work was to screen for sleep potentiated epileptiform discharges in children with language dysfunction.
* To evaluate effect of treatment of these epileptiform discharges on Language dysfunction improvement .

Patients and methods :

* Type of Study: Observational longitudinal study.
* Study Period: From February 2020 till November 2021 .
* Study Population: Patients was recruited from the Pediatric Neurology Clinic, Pediatric Outpatient Clinic, Phoniatrics Outpatient Clinic and the Inpatient Neurology ward at the Ain Shams University Children hospital, Cairo, Egypt.
* Inclusion Criteria: The study was conducted on Children with :

  * Language delay (their language age is below their chronological age ),or Language regression (any convincing report of loss of previously acquired language skills, whether or not prior language development was reported as normal or delayed) (Meilleur et al., 2009)
  * Age from 3 to 10 years old.
* Exclusion Criteria:

  * Patients with hearing problems.
  * Patients whose language delay can be explained by organic disease (e.g. post Hypoxic ischemic encephalopathy, known inborn error of metabolism - whether this language delay is isolated or occurring in the context of global developmental delay).
  * Patients with mental delay.
  * Patients with autism spectrum disorder ( according to DSM-5 standardized criteria, 2013)
  * Enviromentally deprived patients.
* Sampling Method: Consecutive random sampling .
* Sample Size: 93 patients with delayed or regressed language development. (Using PASS 11 program for sample size calculation and according to Nasr et al. (2001), the expected frequency of children with epileptiform discharges =15-60%, assuming that frequency in study population =40%±10%, sample size of 93 children can detect this frequency at 95% confidence level).
* Ethical Considerations: A written informed consent was taken from the parents or legal guardians before enrolment, after fully explaining to them the nature of the study.

The approval of the Research Ethics Committee at Ain Shams University was obtained ( M.D 4312020 ) .

* Study Procedures:

  1. Full history taking:

     * Detailed developmental history.
     * Family history of same condition.
     * History of seizures.
  2. Clinical examination including:

     * General examination.
     * Full neurological examination.
     * Vocal tract examination.
  3. Clinical diagnostic aids :

     * IQ assessment by rapid screening test of Stanford Binet 5th version (Hanoura, 2002).
     * Assessment of language age by modified pre-school language screening test - the Arabic version (Abou-Hassiba, 2011).
  4. Investigations:

     * MRI of the brain will be done. ((1.5 T) Phillips Achieva and Inginea )
     * Auditory brainstem response (ABR). (GSI Audera will be used for acquiring ABR waveforms).
     * 90 minutes sleep EEG (one full sleep cycle) (using Nicolet REF 515-019000 rev 06, CareFusion, Middletown, WI 53562, USA) and placing electrodes by 10-20 placement system.

     Patients whose EEG showed epileptogenic activity ,received treatment and a follow up EEG and Assessment of language age by modified pre-school language screening test - the Arabic version will be done after 6 months.
* Statistical Analysis: Numerical data will be summarized using mean and standard deviations or medians and inter quartile ranges. Qualitative data will be presented as count and percentage, p-value <0.005 will be considered significant.
* Statistical Package: Statistical analysis will be performed with statistical package for social science (SPSS)version 23.0 (SPSS Inc., Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* o Language delay (their language age is below their chronological age ),or Language regression (any convincing report of loss of previously acquired language skills, whether or not prior language development was reported as normal or delayed) (Meilleur et al., 2009)

  * Age from 3 to 10 years old.

Exclusion Criteria:

* o Patients with hearing problems.

  * Patients whose language delay can be explained by organic disease (e.g. post Hypoxic ischemic encephalopathy, known inborn error of metabolism - whether this language delay is isolated or occurring in the context of global developmental delay).
  * Patients with mental delay.
  * Patients with autism spectrum disorder ( according to DSM-5 standardized criteria, 2013)
  * Enviromentally deprived patients.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
language age of the patient | 6 months
  we follow up language age of the patient after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Omnia Alaa Mahsoub, Cairo, Egypt